CLINICAL TRIAL: NCT01059175
Title: Dual-Site LV Pacing in CRT Non Responders Multicenter Randomized V3 Trial
Brief Title: Dual-Site LV Pacing in CRT Non Responders: Multicenter Randomized Trial
Acronym: V3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Collaborators: Medtronic (Industry); FRANCE (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Medtronic
Record Dates: First submitted 2010-01-26; First posted 2010-01-29 (Estimated); Results first posted 2017-04-21 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2017-04

CONDITIONS: Heart Failure
Keywords: Heart failure; Cardiac resynchronization therapy; Biventricular stimulation; Multisite stimulation; Non responders
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CRT With Dual Site LV Pacing (Experimental): Cardiac resynchronization therapy with the addition of a second LV lead. Positioning of a pacing lead in a cardiac vein should be considered first. An epicardial lead will be used if the implant of an endocardial lead is impossible or previously failed.
  Interventions: Device: Additional Endocardial or Epicardial LV Lead; Device: CRT-P or CRT-D
- Standard CRT (Active Comparator): Conventional cardiac resynchronization therapy. Patients in this arm will keep their CRT system unchanged.
  Interventions: Device: CRT-P or CRT-D

INTERVENTIONS:
Device: Additional Endocardial or Epicardial LV Lead — Addition of a second left ventricular endocardial or epicardial lead
  Arms: CRT With Dual Site LV Pacing
Device: CRT-P or CRT-D — Implantable Cardiac Resynchronization Therapy Pacemaker (CRT-P) or Defibrillator (CRT-D) Device

SUMMARY:
Cardiac resynchronization therapy (CRT) is an effective treatment of heart failure (HF) refractory to optimal medical management, in presence of a depressed left ventricular (LV) ejection fraction and a wide QRS complex. It is mainly limited by a high proportion of non-responders. Attempts have been made, in small studies, to increase the number of stimulation sites in order to optimize the resynchronization therapy. V3 is a planned multicenter, randomized trial whose objective is to evaluate the clinical benefit conferred by the addition of a second endocardial or epicardial LV lead in non-responders after at least 6 months of standard biventricular stimulation.

The V3 trial will examine the clinical benefit conferred by the addition of a second LV lead in non-responders compared to standard CRT.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 years
* Recipient of a CRT-P or CRT-D system for greater than 6 for standard indications, including LV ejection fraction greater than 35 percent and New York Heart Association (NYHA) functional class III or IV
* Optimized biventricular stimulation and medical therapy since implantation of the system
* Presence of sinus rhythm, or atrial fibrillation with spontaneous or induced complete atrio-ventricular block
* Greater than 93 percent LV stimulation since the last device interrogation, with a LV capture threshold less than 5.0 Volts/0.5 milliseconds
* Unchanged or worsened clinical status by CRT, according to the HF composite endpoint described by M. Packer, in absence of a reversible cause
* Signature of a written, informed consent to participate in the trial

Exclusion Criteria:

* LV lead location in the great cardiac vein
* Life-expectancy less than 1 year due to concomitant, non-cardiovascular disorders
* Chronic renal dialysis
* Concomitant disorder which might interfere with the results of the V3 trial
* Blood systolic pressure greater than 180 millimeters of mercury (mmHg) or diastolic pressure greater than 95 mmHg despite optimal medical management
* History of stroke, myocardial infarction or unstable angina pectoris within the last 3 months
* Presence of correctible valvular disease
* Subject unable to attend follow-up at the investigative center or unable, for physical or mental reasons, to comply with the trial's procedures, or to sign the informed consent
* Subject is pregnant
* Subject participates in another research project

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2010-09; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bordachar, MD, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- University hospital Rennes, Rennes, France

REFERENCES:
- [Background] Bordachar P, Alonso C, Anselme F, Boveda S, Defaye P, Garrigue S, Gras D, Klug D, Piot O, Sadoul N, Leclercq C. Addition of a second LV pacing site in CRT nonresponders rationale and design of the multicenter randomized V(3) trial. J Card Fail. 2010 Sep;16(9):709-13. doi: 10.1016/j.cardfail.2010.04.010. Epub 2010 Jun 8. PMID 20797593
- [Derived] Bordachar P, Gras D, Clementy N, Defaye P, Mondoly P, Boveda S, Anselme F, Klug D, Piot O, Sadoul N, Babuty D, Leclercq C. Clinical impact of an additional left ventricular lead in cardiac resynchronization therapy nonresponders: The V3 trial. Heart Rhythm. 2018 Jun;15(6):870-876. doi: 10.1016/j.hrthm.2017.12.028. Epub 2017 Dec 26. PMID 29288035

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CRT With Dual Site LV Pacing | Standard CRT
Started | 43 | 41
Completed | 22 (17 patients deceased 4 additional patients were prematurely exited) | 21 (17 patients deceased 3 patients were prematurely exited)
Not Completed | 21 | 20
Not completed — Death | 17 | 17
Not completed — Adverse Event | 4 | 2
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Population: One patient of the V3 group was not included in the ITT analysis of efficacy results as he did not meet inclusion criteria so 83 pts were analyzed
Groups:
- Total: Total of all reporting groups
Arm/Group | CRT With Dual Site LV Pacing | Standard CRT | Total
Number analyzed (Participants) | 42 | 41 | 83
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.5 (7.7) | 72.2 (7.9) | 71.3 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 11
  Male | 36 | 36 | 72
Patients with ischemic heart disease [Number; unit: participants] | 22 | 24 | 46
Paced QRS duration [Mean (Standard Deviation); unit: milliseconds] | 165 (30.5) | 155 (42.2) | 160 (36.8)
Time from first CRT implant [Mean (Standard Deviation); unit: months] | 43.5 (28.4) | 37.8 (23.7) | 40.6 (26.2)
LVEF % (left ventricle ejection fraction) [Mean (Standard Deviation); unit: percent] | 26.9 (6.0) | 25.9 (7.0) | 26.4 (6.4)
LVEDV (left ventricular end-diastolic volume) [Mean (Standard Deviation); unit: milliliter] | 219 (85.8) | 206 (63.9) | 213 (75.7)
LVESV (left ventricular end-systolic volume) [Mean (Standard Deviation); unit: milliliter] | 154 (61.8) | 149 (58.7) | 151 (59.8)

OUTCOME MEASURES:

1. Primary Outcome: Distribution of "Improved", "Unchanged" and "Worsened" Patients as Defined Per M. Packer's Clinical Composite Score
Description: M. Packer's clinical composite score: patients were classified into 1 of 3 response groups after 12 months follow up : worsened, unchanged, or improved.
  Worsened : if death, hospitalization because of or associated with worsening HF, demonstrated worsening in NYHA functional class at their 12-month visit, or if investigator judges global clinical state has worsened.
  Improved :if they had not worsened and had demonstrated improvement in NYHA functional class, or or if investigator judges global clinical state has improved.
  Unchanged : if none of the previous definition applies.
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | CRT With Dual Site LV Pacing | Standard CRT
Number analyzed (Participants) | 42 | 40
participants
  Improved patients | 11 | 7
  Unchanged patients | 10 | 16
  Worsened patients | 21 | 17

2. Secondary Outcome: Distribution of "Improved", "Unchanged" and "Worsened" Patients as Defined Per M. Packer's Clinical Composite Score
Description: Distribution of "improved", "unchanged" and "worsened" patients as defined per M. Packer's clinical composite score at 24 months post implantation of the second left ventricle lead in comparison to the control group M. Packer's clinical composite score: patients were classified into 1 of 3 response groups after 24 months follow up : worsened, unchanged, or improved.
  Worsened : if death, hospitalization because of or associated with worsening HF, demonstrated worsening in NYHA functional class at their 24-month visit, or if investigator judges global clinical state has worsened.
  Improved :if they had not worsened and had demonstrated improvement in NYHA functional class, or or if investigator judges global clinical state has improved.
  Unchanged : if none of the previous definition applies.
Time Frame: 24 months
Measure: Number; unit: participants
Arm/Group | CRT With Dual Site LV Pacing | Standard CRT
Number analyzed (Participants) | 42 | 40
participants
  Patients improved | 8 | 3
  Patients unchanged | 8 | 12
  Patients worsened | 26 | 25

3. Secondary Outcome: Rate of Adverse Events
Time Frame: 24 months
Measure: Number; unit: participants
Arm/Group | CRT With Dual Site LV Pacing | Standard CRT
Number analyzed (Participants) | 42 | 41
participants
  Patients with at least one AE | 38 | 34
  Patients with at least one severe AE | 33 | 33

4. Secondary Outcome: Changes in 6 Minutes Hall Walk Distance Observed Between the Enrollment and the End of the Study
Description: Changes between baseline and 24months follow up
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | CRT With Dual Site LV Pacing | Standard CRT
Number analyzed (Participants) | 42 | 41
meters | -15.1 (88.0) | 7.5 (96.3)

5. Secondary Outcome: Number of Patients With at Least One Hospitalization Related to Heart Failure Between Randomization and the End of the Study
Time Frame: 24 months
Measure: Number; unit: participants
Arm/Group | CRT With Dual Site LV Pacing | Standard CRT
Number analyzed (Participants) | 42 | 41
participants | 19 | 22

6. Secondary Outcome: Time to First Heart Failure Related Hospitalization
Time Frame: 24 months
Measure: Mean (Standard Error); unit: days
Arm/Group | CRT With Dual Site LV Pacing | Standard CRT
Number analyzed (Participants) | 42 | 41
days | 357.6 (27.17) | 402.4 (41.16)

7. Secondary Outcome: Overall Mortality
Time Frame: 24 months
Measure: Number; unit: participants
Arm/Group | CRT With Dual Site LV Pacing | Standard CRT
Number analyzed (Participants) | 42 | 41
participants | 17 | 17

8. Secondary Outcome: Changes in Echocardiographic Indexes of Left Ventricle Remodeling
Description: Changes between baseline and 24months follow up
Time Frame: 24 months
Population: Number of patients with data available for analysis of this objective
Measure: Mean (Standard Deviation); unit: milliliter
Arm/Group | CRT With Dual Site LV Pacing | Standard CRT
Number analyzed (Participants) | 42 | 41
milliliter
  Changes in LVEDV: number analyzed (Participants) | 19 | 14
  Changes in LVEDV | -16.4 (78.6) | 7.0 (72.1)
  Changes in LVESV: number analyzed (Participants) | 18 | 14
  Changes in LVESV | -14.3 (57.6) | -2.0 (60.6)

9. Secondary Outcome: Changes in Quality of Life Score - Minesota Living With Heart Failure Questionnaire
Description: Changes between baseline and 24 months follow up Minesota Living with Heart Failure Questionnaire: 21 questions - addition of scores from 1 (better) to 5 (worse) for each questions.
Time Frame: 24 months
Population: Number of patients with data available for analysis of this objective
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CRT With Dual Site LV Pacing | Standard CRT
Number analyzed (Participants) | 21 | 21
units on a scale | -7.33 (23.5) | -7.48 (17.2)

ADVERSE EVENTS:
Arm/Group | CRT With Dual Site LV Pacing | Standard CRT
Serious Adverse Events (participants affected / at risk) | 33/42 | 33/41
Other Adverse Events (participants affected / at risk) | 38/42 | 34/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CRT With Dual Site LV Pacing (N=42) | Standard CRT (N=41)
Severe cardiovascular event (Cardiac disorders) | 33 | 33 — Definition as per ISO 14155
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CRT With Dual Site LV Pacing (N=42) | Standard CRT (N=41)
Cardiac AE (Cardiac disorders) | 38 | 34 — Definition as per ISO 14155

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No